CLINICAL TRIAL: NCT07272187
Title: Endoscopic Ultrasound-guided Radiofrequency Ablation for Upper Gastrointestinal Tract Lesions - a Prospective Study
Brief Title: Endoscopic Ultrasound-guided Radiofrequency Ablation for Upper Gastrointestinal Tract Lesions
Acronym: EURAGIL
Status: Recruiting | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Bojan Kovacevic, MD, PhD, Herlev Hospital
Other Study IDs: p-2025-19131
Record Dates: First submitted 2025-11-18; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Insulinoma; Pancreas; MEN1; NETs; Radiofrequency Ablation; Endoscopic Ultrasound (EUS); Conn Syndrome
MeSH Terms: conditions — Insulinoma; Hyperaldosteronism | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing EUS-RFA: The cohort consists of patients with benign pancreatic or adrenal tumors (patients with pNENs, MEN1 and Conns syndrome)
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — Observational study. Patients recieve standard clinical care with routine follow up

SUMMARY:
The goal of this observational study is to evaluate the long-term clinical effectiveness of EUS-RFA and quality of life in patients with pancreatic or adrenal tumors recieving EUS-RFA.

Primary Objectives:

* Clinical effectiveness: To evaluate the proportion of included patients who show doc-umented improvement in their clinical symptoms and biochemical parameters (blood test results) over time.
* Patient satisfaction: To assess patient satisfaction with the procedure and subsequent disease-related quality of life, measured using validated questionnaires.

Secondary Objectives:

* Safety: To determine the proportion of treated patients who experience complications, as defined by the AGREE classification, within 30 days after the procedure.
* Technical success: To assess the proportion of included patients in whom the EUS-RFA procedure can be successfully completed.

Exploratory Objectives:

• To identify factors associated with adverse events and factors related to clinical success or lack there of.

The study is observational. All participant will receive EUS-RFA as part of their standard clinical care.

Participants will:

* Undergo EUS-RFA, in which a fine needle is guided into the tumor using an endo-scope and ultrasound imaging. Radiofrequency energy is applied through the needle to heat and destroy tumor cells while protecting the surrounding tissue.
* Have follow-up visits including blood tests, imaging scans, and clinical evaluations at regular intervals for up to 5 years after treatment.
* Complete validated questionnaires about satisfaction and quality of life.

The study will include approximately 138 patients recruited between 2025 and 2035 from two Danish hospital departments (Herlev and Gentofte Hospital and Rigshospitalet). Data collection will continue until 2040 to assess long-term outcomes.

This study may help determine whether EUS-RFA can serve as a safe and effective alternative to traditional surgery for selected patients with small hormone-producing or benign tumors in the pancreas or adrenal glands, potentially reducing surgical risks and improving recovery and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one or more lesions amendable to undergo EUS-RFA

  * Insulinomas ≤ 25 mm confirmed by a 72-h fasting test, cross-sectional scanning, and a biopsy with low Ki67 index (<10%)
  * Non-functional pNEN lesions between 10-20 mm and growing, confirmed by a biopsy with low Ki67 index (<10%), or larger pNEN lesions in patients who are not candidates for surgical treatment
  * Unilateral APA with benign characteristics on non-contrast enhanced CT located in the left adrenal and confirmed lateralization on AVS

    * Adult habile patients
    * Signed informed consent

Exclusion Criteria:

* Severe multimorbidity (ASA score ≥ IV or ECOG performance score ≥ 4)

  * Uncorrected coagulopathy (INR >1.8 or thrombocyte count < 50 mia/L)
  * Pregnancy
  * Metastatic malignancy with expected remaining life expectancy < 3 years
  * Stenosis in upper GI tract or altered anatomy (e.g. previous gastrectomy) preventing the passage of an echoendoscope

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who meet the above inclusion criteria will be offered participation. Herlev Hospital has a national function, and therefore patients from all regions of Denmark are included.
Sampling Method: Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2040-12-31 (Estimated); Study Completion 2041-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | From enrollment and 5 years forward
  Patient satisfaction measured through validated questionarie SF-36. Scores for each domain range from 0 to 100, with a higher score defining a more favorable state
Clinical efficacy | From enrollment and 5 years forward
  Proportion of included patients with documented biochemical response and symptom improvement, or lesion size decrement/cessation of growth in case of MEN1 patients

SECONDARY OUTCOMES:
Adverse events | From enrollment and 5 years forward
  Proportion of treated patients experiencing AEs as defined by AGREE classification during a 30-day period following the procedure
Technical success | From enrollment and 5 years forward
  Proportion of included patients where EUS-RFA was technically feasible

OTHER OUTCOMES:
Factors associated with adverse events | From enrollment and 5 years forward
  Factors associated with adverse events
Factors associated with clinical success or failure | From enrollment and 5 years forward
  Factors associated with clinical success or failure

CONTACTS AND LOCATIONS:
Overall Officials: Bojan Kovacevic, MD, ph.d., Principal Investigator — Herlev and Gentofte Hospital, Capital Region of Denmark
Locations (1):
- Herlev og Gentofte Hospital, Herlev, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided